CLINICAL TRIAL: NCT03434080
Title: Near-infrared Spectroscopy and Electroencephalography to Assess Cortical Activation During Motor Tasks in Infants and Toddlers With or at High-risk for Cerebral Palsy and Autism Spectrum Disorder Compared to Infants and Toddlers With Typical Development
Brief Title: Near-infrared Spectroscopy and Electroencephalography to Assess Cortical Activation During Motor Tasks in Infants and Toddlers With and Without Cerebral Palsy
Status: Terminated | Type: Observational
Why Stopped: PI Retirement
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 180052; 18-CC-0052
Record Dates: First submitted 2018-02-14; First posted 2018-02-15 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Autism; Cerebral Palsy
Keywords: Infant and Toddler at Risk; Pediatric; Neuroimaging; Brain Function; Voluntary Movement; Natural History
MeSH Terms: conditions — Autistic Disorder; Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Autism Spectrum Disorder: The group with ASD (including all infants less than 3 years of age who are identified as being at high-risk for ASD)
- Cerebral Palsy: The group with CP (including all infants less than 18 months who are identified as being athigh-risk for CP)
- Typical Development toddlers infants: The control group will consist of 50 healthy volunteers with TD

SUMMARY:
Background:

New ways to study the brain as people move include near-infrared spectroscopy (NIRS) and electroencephalography (EEG). NIRS uses laser light shone through the scalp to look at blood flow in the brain which increases with movement. EEG records electrical activity in the brain. Little is known about brain activity while children learn new motor skills. Researchers want to learn more about how small children with and without cerebral palsy use their brain to control their body. This may help them find new ways to help children move better.

Objectives:

To learn more about how infants and young children with and without cerebral palsy use their brain to move their arms and legs.

Eligibility:

Children ages 3 months - 5 years with and without cerebral palsy

Design:

Participants will be screened with:

* Physical exam
* Questions for the parents about the child s health

Participants will have at least 1 study session. Some may have up to 34 (all optional).

In the sessions, participants will do motor tasks along with some or all of the following:

* Light sensors placed on the scalp, held there with a cap or Velcro straps.
* Small metal disks placed on the scalp with a cap or straps, with gel between them.
* Motion capture recording. Balls attached to the arms and legs by stickers, straps, or a garment are tracked by infrared and video cameras.

Motor tasks include reaching, clapping, kicking, and standing.

Participants may be placed in a toy or device that uses a motor to move their limbs.

Participants head size, hair, and skin will be assessed.

Parents will answer questions about their child s typical movements.

...

DETAILED DESCRIPTION:
OBJECTIVE

Portable neural imaging during functional tasks is now possible utilizing noninvasive near-infrared spectroscopy (NIRS) which identifies areas of brain activity by measuring blood flow dynamics and electroencephalography (EEG) which measures electrical activity on the cortical surface. Use of these technologies for studying movement is rapidly increasing; however, investigations in children and those with neurological disorders such as cerebral palsy (CP) or autism spectrum disorder (ASD) are still in the early stages with few reports in the literature. The objectives of this protocol are to systematically compare cortical activation patterns during specified sensorimotor tasks in infants and young children with typical development (TD) to those with and at high-risk for CP and ASD, examine developmental changes in brain activation patterns that underlie the emergence of early functional or dysfunctional motor control and explore the neural and biomechanical effects of different devices that make movement easier for infants and toddlers with CP and ASD. The results are expected to increase knowledge of brain activation patterns across tasks in groups with and without neurological disorders and to suggest potential mechanisms or strategies for future clinical intervention trials.

STUDY POPULATION

The group with CP (including all infants less than 18 months who are identified as being at high-risk for CP) will consist of up to 100 children ages 3 months up to 5 years of age. The group with ASD (including all infants less than 3 years of age who are identified as being at high-risk for ASD) will consist of up to 100 children ages 3 months up to 5 years of age. The control group will consist of up to 100 children with TD within the same age range.

DESIGN

This is an observational study that will include cross-sectional and longitudinal data collection. NIRS and/or EEG responses, and kinematic and/or kinetic, force plate, wearable sensors, and/or electromyography (EMG) recordings will be collected on all participants during the performance of self-initiated motor tasks. Additionally, we will evaluate brain and motor responses to devices that aim to make movement easier for infants and children who may have difficulty initiating or performing these movements without assistance.

OUTCOME MEASURES

Primary outcomes are the magnitude, extent and location of brain activity recorded by NIRS and/or EEG within tasks across subject groups. We will also quantify changes in brain activation across ages (cross-sectional) and time (longitudinal). Secondary outcomes may include motion, force plate, wearable sensors, and EMG data to help interpret task and group differences and measures of motor abilities. The same outcome measures will be compared across ages to examine the development of cortical activation patterns and motor abilities and how these change over time and across groups with and without neurological disorders.

ELIGIBILITY:
* INCLUSION CRITERIA:
* All subjects must be between age 3 months up to 5 years of age.
* A healthy volunteer, or
* A child with or at high risk for CP or ASD:

  * An infant/child with an established diagnosis of CP, or
  * An infant less than 18 months who has been identified by a physician as being at high risk for having CP, or
  * An infant/child with an established diagnosis of ASD or
  * A child less than 3 years of age who has been deemed at high-risk for ASD or developmental delays by a physician, early intervention specialist (enrolled in early intervention services), or other qualified health professional, or
  * A younger sibling to a child diagnosed with ASD

EXCLUSION CRITERIA:

* Has any injury or health condition other than CP or ASD or being at-risk for having CP or ASD that affects the ability to move a body part repetitively for short periods. Examples include spinal cord injury, muscle diseases, congestive heart failure, or recently broken bones. The physician or other qualified health professioinal will discuss the child s health history during the screening to determine if participation is safe.
* Child of investigators and children of subordinates to an investigator
* Has a known genetic disorder that is a direct cause of the developmental delays

Additional exclusion criteria for infants and young children with or at high risk for CP:

* Concurrent use of medicines for muscle tone (e.g., baclofen, trihexyphenedyl, dantrolene sodium, tizanidine, or carbidopa/levodopa).
* Has had surgery involving the musculoskeletal system (bone, joints, tendons, muscles, or neurological system (brain, spinal cord, peripheral nerves) within the past year
* Botulinum toxin injections within the past four months.
* A history of having had a major seizure or now diagnosed as having a seizure disorder and is on medication for seizures (e.g. may have had a mild seizure(s) in the past but is not currently being treated for seizures).
* Chronic respiratory problems that require the use of oxygen.

Additional exclusion criteria for infants and young children with or at high-risk for ASD:

* Has had surgery involving the musculoskeletal system (bone, joints, tendons, muscles, or neurological system (brain, spinal cord, peripheral nerves) within the past year.
* Has uncontrollable seizures (e.g. unable to be managed with medicines or treatment).

Additional exclusion criteria for infants and young children with TD

-Born preterm (defined as less than 36 weeks gestation); or birth weight significantly below normal for gestational age (SGA- small for

gestational age).

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 1. patient diagnosed with Autism or infant at high risk ASD. 2. patient diagnosed with CP or infant under 18 months for being at high risk with CP. 3. Typical Development kids (TD).
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2018-05-16 (Actual); Primary Completion 2025-08-21 (Actual); Study Completion 2025-08-21 (Actual)

PRIMARY OUTCOMES:
Magnitude, extent and location of brain activity recorded by NIRS and/or EEG within tasks across subject groups. We will also quantify changes in brain activation across ages (cross-sectional) and time (longitudinal). | each visit
  Data from each of the techniques will be compared across subjects group.

SECONDARY OUTCOMES:
Secondary outcomes include motion and EMG data to help interpret task and group differences and measures of motor abilities. The same outcome measures will be compared across ages to examine the development of cortical activation patterns and mo... | Each Visit
  Outcome measures quantified the type and extent of movement.

CONTACTS AND LOCATIONS:
Overall Officials: Diane L Damiano, Ph.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
Protocol is silent in IPD sharing.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2018-CC-0052.html